CLINICAL TRIAL: NCT00797667
Title: A Phase IIa, Multicenter, Randomized, Placebo-controlled Clinical Trial to Study the Safety and Efficacy of MK0974 for Migraine Prophylaxis in Patients With Episodic Migraine
Brief Title: MK0974 (Telcagepant) for Migraine Prophylaxis in Patients With Episodic Migraine (0974-049)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated based on a recommendation of the DSMB following the identification of two patients with significant elevations in serum transaminases
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0974-049; 2008_591
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telcagepant 140 mg (Experimental): Participants receive one telcagepant 140 mg tablet and one 280 mg telcagepant placebo, orally, twice daily for 12 weeks
  Interventions: Drug: Telcagepant 140 mg; Drug: 280 mg telcagepant placebo
- Telcagepant 280 mg (Experimental): Participants receive one telcagepant 280 mg tablet and one 140 mg telcagepant placebo, orally, twice daily for 12 weeks
  Interventions: Drug: Telcagepant 280 mg; Drug: 140 mg telcagepant placebo
- Placebo (Placebo Comparator): Participants receive one 140 mg telcagepant placebo and one 280 mg telcagepant placebo, orally, twice daily for 12 weeks
  Interventions: Drug: 140 mg telcagepant placebo; Drug: 280 mg telcagepant placebo

INTERVENTIONS:
Drug: Telcagepant 140 mg
  Other Names: MK-0974
  Arms: Telcagepant 140 mg
Drug: Telcagepant 280 mg
  Other Names: MK-0974
  Arms: Telcagepant 280 mg
Drug: 140 mg telcagepant placebo
  Arms: Placebo; Telcagepant 280 mg
Drug: 280 mg telcagepant placebo
  Arms: Placebo; Telcagepant 140 mg

SUMMARY:
A study to assess the safety and efficacy of MK0974 for preventing migraines in patients with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient has had a history of migraine with or without aura
* Patient is able to complete study questionnaire(s) and paper diary

Exclusion Criteria:

* Patient is pregnant or breast-feeding, or is a female expecting to conceive within the projected duration of the study
* Patient has basilar or hemiplegic migraine headache, hepatitis or psychiatric conditions
* Patient was older than 50 years of age at migraine onset
* History of gastric or small intestinal surgery or has a disease that causes malabsorption
* Patient has heart attack, unstable angina, coronary artery bypass surgery or other revascularization procedure, stroke, or transient ischemic attack 3 months before starting the study
* Currently participating or has participated in a study with an investigational compound or device within 30 days of starting the study
* Currently participating in a study with MK-0974 or MK-3207

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2008-11-12 (Actual); Primary Completion 2009-05-20 (Actual); Study Completion 2009-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ho TW, Connor KM, Zhang Y, Pearlman E, Koppenhaver J, Fan X, Lines C, Edvinsson L, Goadsby PJ, Michelson D. Randomized controlled trial of the CGRP receptor antagonist telcagepant for migraine prevention. Neurology. 2014 Sep 9;83(11):958-66. doi: 10.1212/WNL.0000000000000771. Epub 2014 Aug 8. PMID 25107879
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-049&kw=0974-049&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Started | 265 | 264 | 131
Treated | 263 | 263 | 130
Completed | 5 | 5 | 4
Not Completed | 260 | 259 | 127
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 8 | 12 | 2
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Pregnancy | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 7 | 0
Not completed — Study Terminated by Sponsor | 217 | 216 | 115
Not completed — Withdrawal by Subject | 9 | 14 | 2
Not completed — Adverse Event | 19 | 8 | 8

BASELINE CHARACTERISTICS:
Population: All enrolled participants who recieved at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo | Total
Number analyzed (Participants) | 263 | 263 | 130 | 656
Age, Customized [Number; unit: Participants]
  < 20 years | 2 | 3 | 2 | 7
  20-29 years | 54 | 47 | 17 | 118
  30-39 years | 52 | 70 | 43 | 165
  40-49 years | 81 | 80 | 32 | 193
  50-59 years | 66 | 50 | 30 | 146
  60-64 years | 7 | 10 | 2 | 19
  >=65 years | 1 | 3 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 216 | 112 | 551
  Male | 40 | 47 | 18 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Headache Days
Description: Participants entered information about the number of migraine headaches, symptoms, headache pain duration and severity, use of medication, and side effects into a diary each evening just before going to bed. This information was used to determine the mean monthly headache days; a headache day was defined as any day in which a qualified headache (>=30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset was considered an occurrence of multiple distinct headache days. Mean monthly rate was adjusted to 28 days.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS), which included all randomized patients who took at least one dose of study medication and had at least one post-randomization efficacy measurement.
Measure: Mean (95% Confidence Interval); unit: Days per month
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 248 | 247 | 125
Days per month | -3.4 [-3.9 to -2.8] | -3.6 [-4.1 to -3.1] | -2.4 [-3.2 to -1.7]

2. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days
Description: Participants entered information about the number of migraine headaches, symptoms, headache pain duration and severity, use of medication, and side effects into a diary each evening just before going to bed. This information was used to determine the mean monthly migraine days; a migraine day was defined as any day in which a qualified headache( i.e., aura, photophobia, phonophobia, nausea, or vomiting) started, ended, or recurred. Migraine pain persisting for more than 1 calendar day after initial onset was considered an occurrence of multiple distinct migraine days. Mean monthly rate was adjusted to 28 days.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days per month
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 248 | 247 | 125
Days per month | -3.0 [-3.5 to -2.5] | -3.4 [-3.9 to -3.0] | -2.3 [-3.0 to -1.6]

3. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction in Mean Monthly Headache Days
Description: Participants entered information about the number of migraine headaches, symptoms, headache pain duration and severity, use of medication, and side effects into a diary each evening just before going to bed. This information was used to determine the mean monthly headache days; a headache day was defined as any day in which a qualified headache (>=30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset was considered an occurrence of multiple distinct headache days. Mean monthly rate was adjusted to 28 days. The percentage of participants who had at least a 50% reduction in mean monthly headache days during the 12 weeks treatment period was summarized
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 248 | 247 | 125
Percentage of Participants | 36.7 [30.68 to 43.02] | 40.1 [33.92 to 46.48] | 25.6 [18.22 to 34.18]

4. Secondary Outcome: Change From Baseline in the Mean Monthly Migraine Attacks
Description: Participants entered information about the number of migraine headaches, symptoms, headache pain duration and severity, use of medication, and side effects into a diary each evening just before going to bed. This information was used to determine the mean monthly migraine days; a migraine day was defined as any day in which a qualified headache was accompanied with associated symptoms.( i.e., aura, photophobia, phonophobia, nausea, or vomiting) started, ended, or recurred. A migraine attack was defined as any migraine headache that occurs within 2 consecutive calendar days. Pain persisting for more than 2 days after its initial onset was considered a new, distinct migraine attack. The number of migraine attacks that occurred per month was calculated. Mean monthly rate was adjusted to 28 days.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: attacks per month
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 248 | 247 | 125
attacks per month | -2.1 [-2.4 to -1.7] | -2.5 [-2.8 to -2.2] | -1.7 [-2.2 to -1.2]

5. Secondary Outcome: Change From Baseline in the Mean Number of Days Per Month Requiring Rescue Medication
Description: Participants completed a diary each evening just before going to bed. Information recorded included: date of assessment, administration of study medication, medication to treat breakthrough migraines and other headaches, associated symptoms, duration of headache pain, headache severity, and side effects. Participants use of medication to treat a breakthrough migraine/headache was considered rescue medication. The number of days per month requiring rescue medication was calculated.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Days per month
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 248 | 248 | 125
Days per month | -3.0 [-3.5 to -2.5] | -3.2 [-3.7 to -2.8] | -1.7 [-2.4 to -1.0]

6. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event
Description: Participants were assessed throughout the study for adverse events and recorded adverse events in a daily dairy. An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an adverse event.
Time Frame: up to 14 days after last dose of study drug (up to 12 weeks)
Population: All Patients as Treated, which consisted of all participants who received at least 1 dose of study drug and were included in the treatment arm corresponding to the study treatment actually received. If participants took incorrect or mixed study treatment they were included in treatment arm corresponding to the highest dose they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 263 | 265 | 128
Percentage of Participants | 52.5 | 54.0 | 57.8

7. Primary Outcome: Percentage of Participants Who Had Study Drug Discontinued During the Study Due to an Adverse Event
Description: Participants were assessed throughout the study for adverse events and recorded adverse events in a daily dairy. An adverse event was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an adverse event. The percentage of participants who discontinued study was summarized.
Time Frame: up to 12 weeks
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Telcagepant 140 mg | Telcagepant 280 mg | Placebo
Number analyzed (Participants) | 263 | 265 | 128
Percentage of Participants | 8.0 | 3.0 | 7.8

ADVERSE EVENTS:
Time Frame: up to 14 days after last dose of study drug (up to 12 weeks)
Description: All Patients as Treated, which consisted of all participants who received at least 1 dose of study drug and were included in the treatment arm corresponding to the study treatment actually received. If participants took incorrect or mixed study treatment they were included in treatment arm corresponding to the highest dose they actually received.
Groups:
- MK-0974 140 mg: Participants receive one telcagepant 140 mg tablet and one 280 mg telcagepant placebo, orally, twice daily for 12 weeks
- MK-0974 280 mg: Participants receive one telcagepant 280 mg tablet and one 140 mg telcagepant placebo, orally, twice daily for 12 weeks
Arm/Group | MK-0974 140 mg | MK-0974 280 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/263 | 3/265 | 1/128
Other Adverse Events (participants affected / at risk) | 61/263 | 73/265 | 30/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0974 140 mg (N=263) | MK-0974 280 mg (N=265) | Placebo (N=128)
Colonic atony (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0974 140 mg (N=263) | MK-0974 280 mg (N=265) | Placebo (N=128)
Diarrhoea (Gastrointestinal disorders) | 21 (26) | 9 (9) | 6 (6)
Nausea (Gastrointestinal disorders) | 31 (42) | 37 (42) | 7 (10)
Fatigue (General disorders) | 11 (11) | 14 (14) | 11 (12)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 9 (10) | 12 (13)
Dizziness (Nervous system disorders) | 15 (26) | 16 (19) | 7 (13)
Insomnia (Psychiatric disorders) | 6 (8) | 6 (6) | 7 (7)

LIMITATIONS AND CAVEATS:
Based on a recommendation from the external Data Safety Monitoring Board (DSMB), a decision to terminate the trial was made on 26-Mar-2009.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.